CLINICAL TRIAL: NCT04579952
Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Exercise Versus Sham tDCS and Exercise on Pain Control in Chronic Painful Total Knee Arthroplasty (TKA)
Brief Title: Effects of Transcranial Direct Current Stimulation on Pain Control in Chronic Painful Total Knee Arthroplasty
Acronym: TSEF-PTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 687-2019-Disp-IOR
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pain, Chronic
Keywords: Total knee arthroplasty; Chronic pain; Transcranial direct current stimulation
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Single center, double blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant blinding: sham tDCS is provided by a 15 second activation (to perform initial sensation) and then no stimulation in the same areas and with the same cadence of the real tDCS.
  Outcomes assessor blinding: the assessor who evaluates the participants doesn't know if the tDCS or sham tDCS will be or were performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The IG will receive a 20 minute program of active tDCS (2mA intensity, anode placed on primary motor cortex controlateral to the TKA, cathode placed on controlateral supraorbital region) followed by a 30 minute exercise program, 5 days a week, for 2 consecutive weeks.
  Interventions: Device: transcranial Direct Current Stimulation
- Control Group (Placebo Comparator): The CG will receive a 20 minute program of sham tDCS (15 seconds of activation and then no stimulation, same position of IG) followed by the same 30 minute exercise program, 5 days a week, for 2 consecutive weeks.
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — The current stimulation will be applied using 35 squares cm wide sponge electrodes

SUMMARY:
The TSEF-PTG study aims to evaluate the effects of transcranial Direct Current Stimulation (tDCS) and exercise versus sham tDCS (placebo) and exercise on pain control in chronic painful total knee arthroplasty (TKA) patients.

DETAILED DESCRIPTION:
The TSEF-PTG study is a single center, double blinded randomized controlled trial.

The aim is to evaluate the effects of a tDCS stimulation and exercise vs sham tDCS and exercise on pain control in chronic (lasting more than 3 months from the intervention) painful total knee arthroplasty (TKA) patients.

The participants will be randomized in two groups: intervention group (IG) and control group (CG).

The IG will receive a 20 minute program of active tDCS (2mA intensity, anode placed on primary motor cortex controlateral to the TKA, cathode placed on controlateral supraorbital region) followed by a 30 minute exercise program, 5 days a week, for 2 consecutive weeks.

The CG will receive a 20 minute program of sham tDCS (15 seconds of activation and then no stimulation, same position of IG) followed by the same 30 minute exercise program, 5 days a week, for 2 consecutive weeks.

The participants will be evaluated at T0 (enrolling), T1 (at the end of the program), T2 (at 1 month from the end of the program) and T3 (at 3 months from the end of the program).

The primary outcome is the variation of pain intensity, the secondary outcomes are the variation of knee function and of the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* able to independently walk (with or without walk aids)
* chronic painful TKA (more than 3 months)
* Visual Analogic Scale for pain more than 3/10
* No cognitive impairments (MMSE>24 or =24/30)

Exclusion Criteria:

* intracranial metal devices, pacemakers or any implantable devices
* cutaneous abnormalities on the stimulation sites
* epilepsy (past or present)
* neurological or psychiatric pathologies
* cognitive impairment (MMSE<24/30)
* no opioids abuse (past or present)
* severe cardiopulmonary, renal or hepatic pathologies
* pregnancy
* known present TKA complications (e.g. infections, mobilization, etc...)
* pain therapy modifications in the last 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change of pain intensity | Enrollment (T0), at 2 weeks (T1), at 1 month (T2), at 3 months (T3)
  Visual Analogic Scale (VAS) From 0 (no pain) to 10 (worst pain). Higher the score, worse the outcome.
Change of pain characteristics | Enrollment (T0), at 2 weeks (T1), at 1 month (T2), at 3 months (T3)
  Pain detect questionnaire (PD-Q) From 0 to 38. 0-12 more than 75% chance of presence of nociceptive pain. 13-18 uncertain neuropathic pain presence. 19-38 more than 90% chance of neuropathic pain presence. Higher the score, higher the chance of neuropathic pain presence versus nociceptive pain presence.
Change of neuropathic pain presence | Enrollment (T0), at 2 weeks (T1), at 1 month (T2), at 3 months (T3)
  Douleur Neuropathique 4 (DN4) scale From 0 to 10. If score > 4: neuropathic pain presence. Higher the score, higher the chance of neuropathic pain presence.

SECONDARY OUTCOMES:
Knee function | Enrollment (T0), at 2 weeks (T1), at 1 month (T2), at 3 months (T3)
  Knee Society Score (KSS) Knee score 0-100, higher the score, better the characteristics of the knee. Function score 0-100, if score <60 poor function, if score 60-69 fair function, if score 70-79 good function, if score 80-100 excellent function. Higher the score better the knee function.
QoL: Short Form 12 | Enrollment (T0), at 2 weeks (T1), at 1 month (T2), at 3 months (T3)
  Short Form 12

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bardelli, MD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim DH, Pearson-Chauhan KM, McCarthy RJ, Buvanendran A. Predictive Factors for Developing Chronic Pain After Total Knee Arthroplasty. J Arthroplasty. 2018 Nov;33(11):3372-3378. doi: 10.1016/j.arth.2018.07.028. Epub 2018 Aug 4. PMID 30143334
- [Background] Liu SS, Buvanendran A, Rathmell JP, Sawhney M, Bae JJ, Moric M, Perros S, Pope AJ, Poultsides L, Della Valle CJ, Shin NS, McCartney CJ, Ma Y, Shah M, Wood MJ, Manion SC, Sculco TP. A cross-sectional survey on prevalence and risk factors for persistent postsurgical pain 1 year after total hip and knee replacement. Reg Anesth Pain Med. 2012 Jul-Aug;37(4):415-22. doi: 10.1097/AAP.0b013e318251b688. PMID 22660483
- [Background] Scott CE, Howie CR, MacDonald D, Biant LC. Predicting dissatisfaction following total knee replacement: a prospective study of 1217 patients. J Bone Joint Surg Br. 2010 Sep;92(9):1253-8. doi: 10.1302/0301-620X.92B9.24394. PMID 20798443
- [Background] Baert IA, Lluch E, Mulder T, Nijs J, Noten S, Meeus M. Does pre-surgical central modulation of pain influence outcome after total knee replacement? A systematic review. Osteoarthritis Cartilage. 2016 Feb;24(2):213-23. doi: 10.1016/j.joca.2015.09.002. Epub 2015 Sep 14. PMID 26382109
- [Background] Phillips JR, Hopwood B, Stroud R, Dieppe PA, Toms AD. The characterisation of unexplained pain after knee replacement. Br J Pain. 2017 Nov;11(4):203-209. doi: 10.1177/2049463717719774. Epub 2017 Jul 31. PMID 29123665
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Mar 16;3(3):CD008208. doi: 10.1002/14651858.CD008208.pub4. PMID 29547226
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Nikolin S, Huggins C, Martin D, Alonzo A, Loo CK. Safety of repeated sessions of transcranial direct current stimulation: A systematic review. Brain Stimul. 2018 Mar-Apr;11(2):278-288. doi: 10.1016/j.brs.2017.10.020. Epub 2017 Oct 31. PMID 29169814
- [Result] Khedr EM, Sharkawy ESA, Attia AMA, Ibrahim Osman NM, Sayed ZM. Role of transcranial direct current stimulation on reduction of postsurgical opioid consumption and pain in total knee arthroplasty: Double randomized clinical trial. Eur J Pain. 2017 Sep;21(8):1355-1365. doi: 10.1002/ejp.1034. Epub 2017 Apr 25. PMID 28440034
- [Result] Borckardt JJ, Reeves ST, Robinson SM, May JT, Epperson TI, Gunselman RJ, Schutte HD, Demos HA, Madan A, Fredrich S, George MS. Transcranial direct current stimulation (tDCS) reduces postsurgical opioid consumption in total knee arthroplasty (TKA). Clin J Pain. 2013 Nov;29(11):925-8. doi: 10.1097/AJP.0b013e31827e32be. PMID 23370085
- [Result] Chang WJ, Bennell KL, Hodges PW, Hinman RS, Young CL, Buscemi V, Liston MB, Schabrun SM. Addition of transcranial direct current stimulation to quadriceps strengthening exercise in knee osteoarthritis: A pilot randomised controlled trial. PLoS One. 2017 Jun 30;12(6):e0180328. doi: 10.1371/journal.pone.0180328. eCollection 2017. PMID 28665989
- [Result] Wylde V, Dennis J, Gooberman-Hill R, Beswick AD. Effectiveness of postdischarge interventions for reducing the severity of chronic pain after total knee replacement: systematic review of randomised controlled trials. BMJ Open. 2018 Feb 28;8(2):e020368. doi: 10.1136/bmjopen-2017-020368. PMID 29490967
- [Result] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357